CLINICAL TRIAL: NCT05458648
Title: A Prospective Single Center Pilot Study Using the ECGenius System to Collect Electrogram Data to Test an Ablation Impact Algorithm
Brief Title: Single Center Pilot Study Using the ECGenius System to Collect Electrogram Data to Test an Ablation Impact Algorithm
Status: Completed | Type: Observational
Sponsor: CathVision ApS (Industry)
Responsible Party: Sponsor
Other Study IDs: CVAR-00001-A
Record Dates: First submitted 2022-06-17; First posted 2022-07-14 (Actual); Results first posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Persistent Atrial Fibrillation; Cardiac Arrhythmia
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Persistent AF Arm: Patients undergoing cardiac ablation for the treatment of persistent atrial fibrillation
  Interventions: Procedure: Cardiac Ablation for the treatment of persistent Atrial Fibrillation

INTERVENTIONS:
Procedure: Cardiac Ablation for the treatment of persistent Atrial Fibrillation — Patients participating in the study will undergo a cardiac ablation for the treatment of persistent atrial fibrillation.

SUMMARY:
To acquire, amplify, digitize, and record atrial intracardiac electrophysiology signals during cardiac electrophysiology studies for the treatment of persistent atrial fibrillation and to use the recorded data to test the performance of an signal complexity visualization algorithm.

DETAILED DESCRIPTION:
A prospective, single-center, pilot study using the CathVision ECGenius® system and the Ablation Impact Analyzer software in radiofrequency (RF) ablation procedures.

Subjects with persistent atrial fibrillation who are indicated to undergo an RF ablation to treat persistent AF may be enrolled in the Study.

Intracardiac signals will be passively recorded using the investigational ECGenius® System in parallel with the commercial (FDA Approved) EP Workmate, Abbott Inc. EP recording system. The investigational device will not be used for direct clinical care decisions or therapy.

The CathVision ECGenius system allows physicians and users to record intracardiac electrograms during human electrophysiological studies including treatments for atrial fibrillation and atrial tachycardias. Improvements to the first-generation system are in development and include software features and algorithms for further analysis and description of signals to improve the clinical utility of the recorded signals. These new algorithms and software features require leveraging clinical use data as part of the development and iteration process.

This study will allow the evaluation of algorithms for advanced signal analysis in a low-risk clinical setting by recording raw electrocardiograms during standard of care cardiac mapping and ablation treatments for tachyarrhythmias, specifically atrial tachycardias and atrial fibrillation. The data will be recorded by a conventional market-approved EP recording system and on a parallel investigational CathVision ECGenius system for subsequent offline prototype analysis. Information from the investigational system and algorithms will not be available to the physician during the treatment and will have no diagnostic or therapeutic impact on the clinical case.

The validation of the automated algorithm will be performed offline.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients will meet all of the following inclusion criteria:

1. Patients scheduled for RF ablation indicated by the investigator for the treatment of persistent atrial fibrillation.
2. Male or female ≥ 21 years of age.
3. Able and willing to provide written informed consent prior to any clinical investigation related procedure.

Exclusion Criteria:

Eligible patients will not meet any of the following exclusion criteria:

1. Current participation in another investigational drug or device study that interferes with this study.
2. Patients who, in the opinion of the investigator, are not candidates for this study.
3. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the patient's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.
4. Life expectancy less than 12 month, in the opinion of the Investigator.
5. Patients who are considered part of any vulnerable population.
6. Patient is a prisoner.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients already referred to undergo a cardiac ablation as treatment for persistent atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry Jacob, MD, Principal Investigator — NYU Langone
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 patient was a screen failure (wrong rhythm) after having signed the informed consent.
Period: Overall Study
Arm/Group | Persistent AF Arm
Started | 36
Completed | 34
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Patient presented in atrial flutter | 1

BASELINE CHARACTERISTICS:
Arm/Group | Persistent AF Arm
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (11.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 28
  More than one race | 0
  Unknown or Not Reported | 5
Height [Mean (Standard Deviation); unit: cm] | 175.28 (11.64)

OUTCOME MEASURES:

1. Primary Outcome: Ability to Collect CS Data
Description: Data collected during the study will be used to test a signal complexity visualization algorithm. The primary outcome measure was the ability of the system to achieve this in each patient.
Time Frame: One day - day of procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Persistent AF Arm
Number analyzed (Participants) | 34
Participants | 34

2. Secondary Outcome: Measurement of AF Cycle Length
Description: Data collected during the study will be used to test an AF cycle length algorithm
Time Frame: At the start of the procedure from the insertion of the CS catheter to the first ablation
Population: Baseline AFCL
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Persistent AF Arm
Number analyzed (Participants) | 34
ms | 169.64 (24.27)

ADVERSE EVENTS:
Time Frame: The day of the procedure
Arm/Group | Persistent AF Arm
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 1/34
Other Adverse Events (participants affected / at risk) | 3/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Persistent AF Arm (N=34)
Hemorrhage (Blood and lymphatic system disorders) | 1 (1) — Procedure related groin hemorrhage
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Persistent AF Arm (N=34)
Hypotension (Cardiac disorders) | 1 (1) — Procedure related low blood pressure
Atrial Tachycardia (Cardiac disorders) | 1 (1) — Atrial arrhythmia
Pericardial Effusion (Cardiac disorders) | 1 (1) — Procedure related pericardial effusion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2022-03-18): https://cdn.clinicaltrials.gov/large-docs/48/NCT05458648/Prot_000.pdf